CLINICAL TRIAL: NCT05244928
Title: Team Training and Medication Administration in an Ambulance Service. A Study of a Team Training Interventions' Impact on Medication Administration, Teamwork, and Patient Safety Culture.
Brief Title: Team Training and Medication Administration in an Ambulance Service
Acronym: TEAM-AMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sykehuset Innlandet HF (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 16797830
Record Dates: First submitted 2022-01-19; First posted 2022-02-17 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2024-03

CONDITIONS: Patient Safety; Medication Administration
Keywords: Patient safety; Team training; Medication administration; Ambulance services; Human factors
MeSH Terms: interventions — Patient Safety

STUDY DESIGN:
Intervention Model Description: A quasi-experimental, pre- post design, imply the framework for how the "Team Strategies and Tools to Enhance Performance and Patient Safety®" intervention will be introduced in the two clusters. To ease the logistics need for training and the implementation, two clusters will be formed from seven ambulance stations within the same organization. The order in which the two clusters will undergo the intervention will be randomized. The intervention will be introduced for one cluster in February 2022, and for the other cluster in September 2022.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cluster 1. (Experimental): The clusters will be formed from two ambulance stations (Approximately 50 participants).
  Interventions: Other: The team training program "Team Strategies and Tools to Enhance Performance and Patient Safety®"
- Cluster 2. (Experimental): The clusters will be formed from five ambulance stations (Approximately 70 participants).
  Interventions: Other: The team training program "Team Strategies and Tools to Enhance Performance and Patient Safety®"

INTERVENTIONS:
Other: The team training program "Team Strategies and Tools to Enhance Performance and Patient Safety®" — "Team Strategies and Tools to Enhance Performance and Patient Safety®" is a team training program consisting of an evidence-based set of tools designed to develop teamwork skills with the goal of improving quality in healthcare services and providing safer patient care. In this study, selected tools from the "Team Strategies and Tools to Enhance Performance and Patient Safety®" curriculum have been chosen for implementation over a 4-month period together with a general emphasis on the key principles: communication, leadership, situation monitoring and mutual support. A full day introduction will be held to mark the start of the intervention and each successive month will have a focus on a single key principle with associated tools.
  A quasi-experimental, pre- post design, provides the framework for the intervention of the team training program in two clusters including seven ambulance stations, in total.

SUMMARY:
Medication administration events have the potential to cause patient harm. Frequency of medication administration events in the ambulance services is less known. Effective teamwork has been described as paramount for providing safe and effective patient care in the high-risk ambulance environment. "Team Strategies and Tools to Enhance Performance and Patient Safety®" is an evidence-based team training program released from the Agency for Healthcare Research and Quality.

The aims of the study are: (1) to advance the knowledge of medication administration process in the ambulance services, and (2) to study the impact of a team training program on medication administration events, teamwork, and patient safety culture.

To address the overall aims, the following research objectives will guide the study:

Pre-study: To analyse and validate the psychometric properties of the Norwegian version of the Teamwork Perception Questionnaire for use in an ambulance service.

Studies:

1. To determine the frequency of medication administration events in an ambulance service.
2. To describe the medication administration process in an ambulance service according to the "Systems Engineering Initiative for Patient Safety model".
3. To identify the impact of a team training program on the frequency of medication administration events in an ambulance service.
4. To explore ambulance professionals' experiences of teamwork before and after the implementation of a team training program and their experiences with the program.
5. To compare ambulance professionals' perceptions of teamwork and patient safety culture before and after implementation of a team training program.

Post-study: To study the association between medication administration events and team training and patient safety culture in an ambulance service.

A quasi-experimental, pre- and post-design, provides the framework for the intervention of the team training program in two clusters including seven ambulance stations, in total.

ELIGIBILITY:
Inclusion criteria pre-study

* Ambulance professionals employed in the ambulance services

Exclusion criteria pre-study

* Under 18 years of age

Inclusion criteria study 1 and 3

* EPJs for patients who are transported or treated within the assigned areas
* Patient which receives medication (Oxygen, or clear fluid intravenously, by inhalation, intramuscularly, intraosseous, per os, sublingually, or intranasally)

Exclusion criteria study 1 and 3

* Missing and/or incomplete data.

Inclusion criteria study 2

* Ambulance professionals employed in the ambulance services

Exclusion criteria study 2

* Under 18 years of age
* Student and apprentices

Inclusion criteria study 4 and 5

* Ambulance professionals and apprentices participating in the "Team Strategies and Tools to Enhance Performance and Patient Safety®" intervention

Exclusion criteria study 4 and 5

* Ambulance professionals on long-term leave
* Under 18 years of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Testing the psychometric properties of the Teamwork Perception Questionnaire | 4 weeks
  The questionnaire will be digitally distributed to approximately 500 ambulance personnel in a hospital trust. Each items are scored on a five-point scale. The survey will be carried out for 14 days in February, and 14 days in August 2022.
The perception of patient safety culture and teamwork. | 3 month
  To measure the ambulance personnel's perception of patient safety culture and teamwork, the Prehospital Survey on Patient Safety Culture (five point-scale) and the Teamwork Perception Questionnaire (five point-scale), will be carried out at three times in each cluster (one time before and two times after the intervention)
  In cluster 1, the survey will be carried out for 14 days in January/February 2022, 14 days in June 2022 and 14 days in January 2023.
  In cluster 2, the survey will be carried out for 14 days in August 2022, 14 days in January 2023 and 14 days in August 2023.
The frequency of medication administration in ambulance service | 18 month
  The frequency of medication administration will be assed by a retrospective review of approximately 500 electronic patient journals before the intervention. An interim analysis will be conducted after the this review to determine the final number of necessary review of electronic patient journals after the intervention. The journals will be collected for a 6-month period prior to the intervention and a 12-month period after the end of the intervention in both clusters.
Description of the medication administration process. | 3 month
  Qualitative data from partly participants observations, approximately 10 individual interviews of ambulance professionals and supplemented by local guidelines.
The experiences of teamwork and the team training program before and after the intervention. | 4 days
  Qualitative data from from four focus group interviews before and after the intervention in each cluster.

SECONDARY OUTCOMES:
Association between medication administration, team training and patient safety culture | 21 month
  The study include data from the primary outcome measures 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Hartz, PhD, Study Director — Sykehuset Innlandet HF
Locations (1):
- Innlandet Hospital Trust, Brumunddal, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Myhr K, Ballangrud R, Porthun J, Sollid SJM, Vifladt A. Medication administration errors in a Norwegian ambulance service: a quasi-experimental study on the impact of a team training program. Scand J Trauma Resusc Emerg Med. 2026 Jan 24. doi: 10.1186/s13049-026-01560-1. Online ahead of print. PMID 41580728
- [Derived] Myhr K, Ballangrud R, Aase K, Vifladt A. Ambulance professionals' experiences of teamwork in the context of a team training programme - a qualitative study. BMC Emerg Med. 2024 Jul 2;24(1):108. doi: 10.1186/s12873-024-01018-6. PMID 38956498
- [Derived] Vifladt A, Ballangrud R, Myhr K, Grusd E, Porthun J, Maehlum PA, Aase K, Sollid SJM, Odberg KR. Team training program's impact on medication administration, teamwork and patient safety culture in an ambulance service (TEAM-AMB): a longitudinal multimethod study protocol. BMJ Open. 2023 Jan 20;13(1):e067006. doi: 10.1136/bmjopen-2022-067006. PMID 36669839